CLINICAL TRIAL: NCT04720638
Title: Clinical Performance of Short Fiber Reinforced Flowable Resin Composite Restorations Versus Conventional Resin Composite Restorations in Posterior Teeth (2y Randomized Clinical Trial)
Brief Title: Clinical Performance of Short Fiber Reinforced Flowable Resin Composite Restorations 2y RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Hesham Abd ElAziz, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU-1-2021
Record Dates: First submitted 2021-01-19; First posted 2021-01-22 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Decay, Dental; Caries Class II
Keywords: short fiber reinforced flowable resin composite; Clinical performance; Ever X flow; Randomized clinical study
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short fiber reinforced flowable resin composite restorations (Experimental): (everX Flow, GC Europe) + (Gaenial posterior, GC Europe
  Interventions: Other: Short fiber reinforced flowable resin composite restorations
- Conventional resin composite restoration. (Active Comparator): (Gaenial posterior, GC Europe)
  Interventions: Other: Conventional resin composite restoration

INTERVENTIONS:
Other: Short fiber reinforced flowable resin composite restorations — reinforced flowable resin composite
  Other Names: Ever X Flow
  Arms: Short fiber reinforced flowable resin composite restorations
Other: Conventional resin composite restoration — Microhybrid resin composite
  Other Names: Gaenial posterior, GC Europe
  Arms: Conventional resin composite restoration.

SUMMARY:
Clinical performance of short fiber reinforced flowable resin composite restorations versus conventional resin composite restorations will be tested in posterior teeth (2y randomized clinical trial).

ELIGIBILITY:
Inclusion Criteria:

* Patients with large proximal carious cavities in molars.
* Pulp asymptomatic vital carious upper or lower molars.
* Good oral hygiene.

Exclusion Criteria:

* Presence of signs and symptoms of irreversible pulpitis or pulp necrosis
* Severe medical complications.
* Allergic history concerning methacrylates
* Evidence of parafunctional habits.

Ages: 17 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Clinical performance (Alpha is the best score, bravo, charlie the worst score) | Change from baseline at 6, 12 ,18, 24 months
  Modified USPHS criteria; . Post operative Hypersensitivity
  Secondary caries
  Gross fracture
  Color match
  Cavo-surface marginal discoloration
  Marginal integrity
  Proximal contact

CONTACTS AND LOCATIONS:
Overall Officials: Rawda Hesham, Principal Investigator — Lecturer at faculty of Dentistry- Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No